CLINICAL TRIAL: NCT02813096
Title: Efficacy and Safety Study of Folfox4 Chemotherapy Regimen to Prevent Early Recurrence of Hepatocellular Carcinoma Patients With Portal Vein Tumor Thrombus Following Curative Resection
Brief Title: Study of Folfox4 Chemotherapy Regimen to Prevent Early Postoperative Recurrence for HCC-PVTT Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jiazhou Ye, M.D., Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GuangxiMUJYe
Record Dates: First submitted 2016-06-16; First posted 2016-06-24 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Carcinoma, Hepatocellular
Keywords: HCC; PVTT; Folofox4; Early Recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- folfox4 chemotherapy regimen (Experimental): details in the "Intervention Description"
  Interventions: Drug: folfox4 chemotherapy regimen
- Placebo (Placebo Comparator): details in the "Intervention Description"
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: folfox4 chemotherapy regimen — Folfox regimen:Oxaliplatin 85 mg/m2 in 250 mL 5% glucose solution, IVD (administered as 2-hour infusion) on day 1;leucovorin 200 mg/m2 in 100 mL 0.9% NaCl solution, IVD (administered as 2-hour infusion) on days 1 and 2; 400 mg/m2 5-FU in 20mL 0.9% NaCl solution, IV(administered as follow leucovorin); then 600 mg/m2 5-FU in 100 mL 0.9% NaCl solution (administered as 22-hour continuous infusion) on days 1 and 2 of each 14 days cycle.
  Number of cycles: 4 cycles, or until progression or unacceptable toxicity develops.
  Other Names: F4 chemo
  Arms: folfox4 chemotherapy regimen
Other: Placebo — Placebo regimen:250 mL 5% glucose solution, IVD (administered as 2-hour infusion) on day 1; 100 mL 0.9% NaCl solution, IVD (administered as 2-hour infusion) on days 1 and 2; 20mL 0.9% NaCl solution, IV; then 100 mL 0.9% NaCl solution (administered as 22-hour continuous infusion) on days 1 and 2 of each 14 days cycle.
  Number of cycles: 4 cycles, or until progression or unacceptable toxicity develops.
  Other Names: control
  Arms: Placebo

SUMMARY:
This study is to investigate the efficacy and safety of Folfox4 chemotherapy regimen to prevent early recurrence for hepatocellular carcinoma patients with portal vein tumor thrombus following curative resection

DETAILED DESCRIPTION:
Curative resective is well-accepted as the predominant treatment for hepatocellular carcinoma (HCC) patients. Unfortunately, the long-term prognosis remains poor due to frequent postoperative recurrence, especially in HCC patients with portal vein tumor thrombus (PVTT). When PVTT invades into the portal vein system, tumor cell spreads and distributes along with the portal vein and its branches,thus resulting in intra-hepatic micro-metastasis which contributes to early recurrence for patients following curative resection. Postoperative adjuvant interventions include TACE, antiviral therapy, immunotherapy, local radiotherapy were applied to prevent recurrence. However, the efficacy and safety of these regimens remains unsatisfactory. Thus new therapeutic strategy remains to be investigated. This study is to investigate the efficacy and safety of Folfox4 chemotherapy regimen to prevent early recurrence for HCC patients with PVTT following curative resection.

ELIGIBILITY:
Inclusion Criteria:

* patients undergo curative resection
* HCC with PVTT is confirmed by pathological examination
* patients undergo chemotherapy of Folfox4 regimen
* patients without recurrence within the first month after curative resection
* residual hepatic function is Child-pugh A or B which is capable to tolerate chemotherapy
* patients without other postoperative adjuvant treatments including TACE, radiotherapy, immunotherapy

Exclusion Criteria:

* Multipal intra-hepatic or outra-hepatic tastasis within the first month after curative resection
* patients with residual hepatic function Child-pugh C is not capable to tolerate chemotherapy
* patients undergo postoperative adjuvant treatments except chemotherapy of Folfox4 regimen
* patients with badly chemotherapy complications who can finish the whole Folfox4 treatment course

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
early recurrence | from date of randomization until the first document recurrence from any cause, whichever came first, assessed up to 2 years

SECONDARY OUTCOMES:
overall survival | from date of randomization until the date of death from any cause, whichever came first, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lequn Li, M.D., Study Chair — Cancer Hospital of Guangxi Medical University; Jiazhou Ye, M.D., Principal Investigator — Cancer Hospital of Guangxi Medical University

IPD SHARING:
Plan to Share IPD: Undecided